CLINICAL TRIAL: NCT05385458
Title: Acceptance and Commitment Therapy (ACT) Through Tele-Counselling for Family Caregivers in New Brunswick
Brief Title: Acceptance and Commitment Therapy (ACT) Tele-Counselling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Collaborators: Alzheimer Society of New Brunswick (Unknown); Mount Allison University (Unknown); University of Ottawa (Other); McMaster University (Other); McGill University (Other)
Responsible Party: Principal Investigator, Pamela Durepos, Assistant Professor, University of New Brunswick
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHRC-NBHRF Mental Health
Record Dates: First submitted 2022-03-21; First posted 2022-05-23 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Acceptance and Commitment Therapy; Caregiver Burden; Digital Health; Technology; Mental Health; Psychotherapy; Counselling; Dementia
MeSH Terms: conditions — Caregiver Burden; Psychological Well-Being; Dementia

STUDY DESIGN:
Intervention Model Description: Two group randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: One investigator who will have no contact with participants will generate a randomization sequence. The research assistant who enrols participants in the studies will be blinded to the randomization sequence. They will contact the investigator to be told what group the participant is allocated. It is not possible to mask participants. Investigators will be blinded to groups when assessing and comparing outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Intervention (Experimental): Participants will attend 6-8 individual psychotherapy sessions via telephone, text or videoconference. Sessions will last approximately 1 hour and occur every 3-4 weeks. Participants will be enrolled in the Intervention Group for 18-36 weeks. All sessions will be audio recorded. Participants will also be able to attend all available usual care services such as: support groups, First Link, education classes at the Alzheimer Society. Any services utilized will be documented by Alzheimer Society staff.
  Interventions: Behavioral: ACT Intervention
- Usual Care (Active Comparator): Participants will be enrolled as an Alzheimer Society client. Participants will receive 1 First Link 'check-in' telephone call from a staff member at the time of enrolment. Participants will receive a 2nd 'check-in' First Link telephone call from a staff member 3-4 months following enrolment. Participants will be enrolled in the Usual Care Group 12-16 weeks. Participants will also be able to attend all available usual care services such as: support groups, etc. Any services utilized will be documented by Alzheimer Society staff.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: ACT Intervention — Acceptance and Commitment Therapy
  Arms: ACT Intervention
Other: Usual Care — Usual Care Services
  Arms: Usual Care

SUMMARY:
A randomized 2-group controlled trial will be conducted to explore the potential effect and potential feasibility of a new Acceptance and Commitment Therapy (ACT) tele-counselling program to improve mental health services for family caregivers of persons with dementia in the province of New Brunswick in Canada. The ACT tele-counselling program was launched in January 2021 with the aim of improving access to high quality psychotherapy for family caregivers, particularly in rural areas. A target sample size of 80 participants will be recruited and randomly allocated to either the ACT program or to usual care services. Mixed methods (QUANTITATIVE + qualitative) will be used to evaluate the potential impact of the ACT program compared to usual care on participant's mental health, and to generate recommendations for the expansion and continuation of the program outside of the province.

DETAILED DESCRIPTION:
Family caregivers of persons with dementia have limited access to high quality psychotherapy in NB and across Canada, despite experiencing high levels of burden, depression, anxiety and social isolation. This feasibility pilot study will use a randomized two-group controlled trial design to evaluate the feasibility, acceptability and potential effect of a new Acceptance and Commitment Therapy (ACT) tele-counselling program offered by the Alzheimer Society of NB to family/friend caregivers. The program was launched in February 2021 and requires evaluation to maintain funding and inform implementation practices (i.e., scale-up) into other provinces.

Approximately 80 French/English-speaking adult caregivers of persons living with dementia will be recruited to participate in the study. We anticipate an attrition rate of approximately 25% and aim to retain a sample of 60 (30 participants per group). Participants will be screened for eligibility and those who demonstrate severe anxiety, depression or stress in 2 or more subscales according to the DASS-21 questionnaire will not be eligible to participate in the study and will be enrolled directly to the ACT program at the Alzheimer Society of NB. Eligible participants will be randomly assigned to either a usual care or intervention group.

Usual Care Group: Participants will receive usual care services at the Alzheimer Society including: First Link check-in telephone call once at the beginning of the study and a 2nd phone call 3 months later from an Alzheimer Society staff member. They would also have access to monthly support groups and education classes as they wish. Use of services will be tracked as per usual by the Alzheimer Society over 12 weeks.

Intervention Group: Participants will attend 6-8 individual tele-counselling sessions over 12-24 weeks with the psychotherapist who developed the ACT program at the Alzheimer Society. Sessions will last 45-60 minutes and be delivered in French or English via text, Zoom or telephone using Health Insurance Portability and Accountability Act (HIPAA) compliant technology. Participants will select their preferred mode of delivery for the program. Sessions will include ACT methods such as: identifying presenting concerns, making contact with the present moment, identifying values, accepting the situation and setting boundaries/expectations, and examining thoughts. All sessions will be recorded and 20% randomly selected to be reviewed by a research team member to evaluate intervention fidelity. Participants can refuse to have their session recorded and remain in the study. Participants in the Intervention Group will also have access to Usual Care services.

Participants will complete a pre-post test with outcome measures completed at baseline (T1) and after attending either Usual Care or the ACT program (T2) to assess potential effect. Participants will complete electronic or paper questionnaires (administered and returned via postal mail). Questionnaires have evidence for reliability and validity in French and English and have been used to evaluate ACT effectiveness in family caregivers. Outcome measures will include: Depression, Anxiety and Stress Scale (DASS-21), Acceptance and Action Questionnaire II (AAQ-11), Zarit Caregiver Burden-6 (ZBI-6), and the Engagement in Meaningful Activities Survey (EMAS).

Feasibility and acceptability of the intervention will be evaluated by tracking participant movement (i.e., recruitment, retention, sessions completed). Participants in the Intervention Group will also complete the System Usability Scale (SUS) and the Client Satisfaction Questionnaire (CSQ-8) after completing the Intervention. Telephone or computer interviews lasting 1 hour will be conducted with 10 participants in the Intervention Group to explore perceptions of the intervention, facilitators and barriers. 1 computer or telephone focus group will be conducted with 5-6 staff members of the Alzheimer Society involved in delivery of the program to explore perceptions and recommendations for program implementation and scale-up. Interviews and the focus group will be audio recorded and transcribed.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 19 years old residing in New Brunswick, Canada
* Able to speak and read English or French
* Unpaid, informal caregiver to a person living with dementia (no diagnosis required)
* High level on 2 subscales or less on the Depression, Anxiety and Stress Scale
* Current or previous use of any mental health services

Exclusion Criteria:

* Less than 19 years old or not residing in New Brunswick, Canada
* Unable to speak and read English or French
* Not an unpaid informal caregiver to a person living with dementia
* High level on more than 2 subscales on the Depression, Anxiety and Stress Scale
* Acute mental health disorder such as: schizophrenia or bipolar disorder

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Depression, Anxiety and Stress up to 36 weeks as assessed by the Depression, Anxiety and Stress Scale | Baseline through study completion up to 36 weeks
  The Depression, Anxiety and Stress Scale (DASS-21) scale has 21 items with a 3 point likert scale. Range is 0-189 with higher scores indicating greater symptoms of depression, anxiety and stress.
Change in Baseline Caregiver Burden up to 36 weeks as assessed by the Zarit Burden Index | Baseline through study completion up to 36 weeks
  The Zarit Burden Index (ZBI-12) is a 12 Item questionnaire with 5 point likert scale. Range is 0-48 with higher scores indicating higher symptoms of caregiver burden.
Change in Baseline Caregiver Participation in Meaningful and Fulfilling Activities up to 36 weeks as assessed by the Engagement in Meaningful Activities Scale | Baseline through study completion up to 36 weeks
  The Engagement in Meaningful Activities Scale (EMAS) assesses the alignment between a person's actions/activities in daily life and their personal values. Increasing engagement in meaningful activities is a goal of ACT. This scale has 12 items with 5 point likert scale. Range is 12-72 with higher scores indicating higher (better) engagement in meaningful activities.
Change in Psychological Flexibility and Experiential Avoidance up to 36 weeks as assessed by the Acceptance and Action Questionnaire | Baseline through study completion up to 36 weeks
  The Acceptance and Action Questionnaire (AAQ-II) was developed to evaluate the effectiveness of ACT behavioural therapy, which aims to increase psychological flexibility and decrease experiential avoidance. Psychological flexibility refers to a person's ability to recognize and adapt to situational demands; shift perspectives, thinking or behaviours that reduce personal or social functioning; maintain balance among important life domains; and be aware, open, and committed to behaviors that align with personal values (Kashdan, 2010). The questionnaire includes 7 Items with a 7 point likert scale. Range is 7-49 with lower scores indicating higher (better) psychological flexibility and lower (better) experiential avoidance.

SECONDARY OUTCOMES:
Acceptability of ACT Intervention Technology Used for Remote Delivery up to 36 weeks as assessed by the System Usability Scale | Through study completion up to 36 weeks
  An adapted version of the System Usability Scale (SUS) will be used to asses how acceptable and easy it is for caregivers to use technology (telephone, text, videoconference) to attend the ACT intervention tele-counselling sessions remotely. The scale includes a 10 item scale with 5 point likert scale. Range is 10-50 with higher scores indicating higher acceptability.
Satisfaction with ACT Intervention Delivery, Content and Processes up to 36 weeks as assessed by the Client Satisfaction Questionnaire | Through study completion up to 36 weeks
  The Client Satisfaction Questionnaire (CSQ-8) scale assesses perceptions of the quality of a service or program, whether the service has met expectations and needs, likelihood of recommending the service to others, and perceived effectiveness/helpfulness of the service. The scale includes 8 items with a 4 point likert scale. Range is 8-32 with higher scores indicating higher satisfaction.
Feasibility and Acceptability of Implementing the ACT Intervention as planned through study completion up to 1 year as assessed by recruitment, retention and attrition rates, and participant demographics | Through study completion up to 1 year
  Feasibility and acceptability of the ACT intervention will be assessed through participant tracking and statistical analysis of frequencies and descriptive statistics to understand recruitment, retention and attrition rates, number of tele-counselling sessions completed, and diversity of participant demographics (i.e., gender, geographical area, language spoken, age) recruited and who complete the study.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Durepos, PhD, Principal Investigator — University of New Brunswick
Locations (1):
- Alzheimer Society of New Brunswick, Fredericton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with researchers outside of the study.

REFERENCES:
- [Derived] Durepos P, Ricketts N, Olthuis JV, Gould ON, Boamah SA, McCloskey R, Lanteigne M, Giberson ER, Caverhill K, Pickford K, MacBean C, Kaasalainen S. Acceptance and Commitment Therapy Tele-Counselling Program With Care Partners of Persons Living With Dementia: A Pilot Feasibility RCT. J Appl Gerontol. 2026 Feb;45(2):225-236. doi: 10.1177/07334648251338303. Epub 2025 May 12. PMID 40353485